CLINICAL TRIAL: NCT06653543
Title: Effect of Mulligan Mobilization With Arm Movement on Nerve Conduction Velocity in Patients With Unilateral Cervical Radiculopathy
Brief Title: Effect of Mulligan on Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tawfik Mohamed Tawfik Elgazar, teaching assistant at the department of basic science, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005110
Record Dates: First submitted 2024-09-01; First posted 2024-10-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cairo University
Keywords: mobilization; Mulligan; cervical; radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mulligan group (Experimental): 20 participants recieving conventional therapy in addition to mulligan mobilization with arm movement
  Interventions: Other: Mulligan mobilization with arm movement; Other: conventional therapy of cevical radiculopathy
- control group (Sham Comparator): control group that revieves only the conventional therapy
  Interventions: Other: conventional therapy of cevical radiculopathy

INTERVENTIONS:
Other: Mulligan mobilization with arm movement — mulligan mobilization applied on cervical spine with arm movement
  Arms: mulligan group
Other: conventional therapy of cevical radiculopathy — hot pack for 10 minutes, active ranges of motion (AROMs) with 3 sets of 10 repetitions and isometrics for each movement repeated 20 times with the hold of 6 to 10 seconds in each repetition

SUMMARY:
The goal of this clinical trial is to investigate the effect of Mulligan mobilization with arm movement on nerve conduction velocity in patients with unilateral cervical radiculopathy. The main questions it aims to answer are :

1. Is there a statistical significant effect of mobilization with arm movement on NCV velocity in treatment of cervical radiculopathy ?
2. Is there a statistical significant effect of mobilization with arm movement on pain level in treatment of cervical radiculopathy ?
3. Is there a statistical significant effect of mobilization with arm movement on cervical ROM in treatment of cervical radiculopathy ?
4. Is there a statistical significant effect of mobilization with arm movement on neck disability level in treatment of cervical radiculopathy ?

The course of treatment involves 6 sessions over the course of 3 weeks participants will be divided into 2 groups : Control group : recieves only Conventional treatment Experimental group : recieves Conventional treatment and Mulligan mobilization with arm movement .

DETAILED DESCRIPTION:
the aim of our study is to examine the effect of Mulligan mobilization with arm movement on cervical radiculopathy using nerve conduction studies , in addition to the original measures of previous studies (pain level, cervical ROM and neck disability scale) .

Delimitations :

Inclusion Criteria

Individuals will be enrolled into the study if they are :

* diagnosed with cervical radiculopathy .
* Age group between 20-60 years
* Unilateral radiating pain through the course of median nerve .
* Subject having positive upper limb tension test (ULTT 1)
* either gender male and female
* Subjects who can understand the instructions and are willing to participate in the study.

Exclusion Criteria .

* History of trauma, dislocation and subluxation of upper extremity
* Rheumatoid Arthritis
* Malignancy
* Spinal canal stenosis .
* Cervical instability/Spondylolisthesis
* VBI (Vertebral-Basillar Insufficiency)
* Referred pain in patients with cardiac ischemia
* Cervical or thoracic spine surgeries
* systemic causes like diabetic neuropathy.
* recent fracture or surgery in and around the shoulder
* carpal tunnel syndrome .
* thoracic outlet syndrome .

Outcome measure would include:

A) The primary outcome measure will be NCV velocity, for the median nerve (latency, amplitude, Duration , F-wave and nerve conduction velocity of motor nerve action potentials and sensory nerve action potentials (SNAPs)) .

B) Secondary outcome measures will include:

* Pain intensity, assessed using the Visual Analog Scale (VAS) .
* Functional disability, evaluated using the Neck Disability Index (NDI) .
* Cervical range of motion, measured using a CROM goniometer to assess flexion, extension, lateral flexion, and rotation.
* The course of treatment involves 6 sessions over the course of 3 weeks .
* pre-treatment for both groups :

  1. affected nerve conduction velocity will be measured using nerve conduction study .
  2. neck disability level will be measured using neck disability index .
  3. cervical ROM measurement will be taken in all directions using CROM goniometer .
  4. pain will be assessed using Visual analog scale .

participants will be divided into 2 groups :

Group A- Control group:

During each session : only Conventional treatment will be provided , includes : hot pack for 10 minutes, active ranges of motion (AROMs) with 3 sets of 10 repetitions and isometrics for each movement repeated 20 times with the hold of 6 to 10 seconds in each repetition.

Group B- Experimental group- Mulligan mobilization group:

* During each session :

  1. Conventional treatment will be provided .
  2. Mulligan mobilization will be applied in the form of : sustained passive accessory joint mobilization to a specific spinal vertebra level while simultaneously guiding the patient through an active, pain-free movement pattern involving the affected limb :
* Patient position : Sitting upright on chair
* Therapist position : Standing behind the patient .
* Hand placement : Approach the desired level of spinous process from medial aspect of the thumb of one hand, which may be reinforced by the index finger of the other hand.
* Mobilization Pure transverse glide is performed from affected to unaffected side. While the glide is sustained, patient performs the offending movements (flexion/abduction/horizontal adduction/horizontal abduction)

ELIGIBILITY:
Inclusion Criteria:

* • diagnosed with cervical radiculopathy .

  * Age group between 20-60 years
  * Unilateral radiating pain through the course of median nerve .
  * Subject having positive upper limb tension test (ULTT 1)
  * either gender male and female
  * Subjects who can understand the instructions and are willing to participate in the study.

Exclusion Criteria:

* • History of trauma, dislocation and subluxation of upper extremity

  * Rheumatoid Arthritis
  * Malignancy
  * Spinal canal stenosis .
  * Cervical instability/Spondylolisthesis
  * VBI (Vertebral-Basillar Insufficiency)
  * Referred pain in patients with cardiac ischemia
  * Cervical or thoracic spine surgeries .
  * systemic causes like diabetic neuropathy .
  * recent fracture or surgery in and around the shoulder .
  * carpal tunnel syndrome .
  * thoracic outlet syndrome .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
median nerve conduction study | 2 weeks
  using nerve conduction studies to measure the median nerve (latency, amplitude, Duration , F-wave and nerve conduction velocity of motor nerve action potentials and sensory nerve action potentials ) .

SECONDARY OUTCOMES:
cervical range of motion | 2 weeks
  using cervical CROM device to measure the cervical ROM in all 3 planes
pain | 2 weeks
  using visual analogue scale for the pain intensity .. where no pain or discomfort(0) , while the severest pain (10) .. the more the pain , the more the points on the scale
neck disability level | 2 weeks
  using neck disability index questionnaire consists of 10 items, where each item is scored on a scale of 0 to 5, with 0 indicating no disability and 5 indicating complete disability
  * The total score ranges from 0 to 50.
  * Higher scores indicate greater disability and impairment, while lower scores indicate less disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El-Sheikh university, Kafr El-Sheikh Governorate, Kafr el-Sheikh Governorate, Egypt